CLINICAL TRIAL: NCT05698992
Title: Rehabilitation and Recovery for Persons with Esophageal or Gastric Cancer - a Clinical Trial Evaluating and Implementing a Model for Evidence-based Cancer Rehabilitation
Brief Title: Rehabilitation and Recovery for Persons with Esophageal or Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Marlene Malmström, Associate professor, Region Skane
Other Study IDs: Esophageal/gastric cancerrehab
Record Dates: First submitted 2022-12-02; First posted 2023-01-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Cancer; Esophageal Neoplasms; Gastric Cancer; Stomach Neoplasm
Keywords: Cancer rehabilitation; Recovery
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental group: Patients over 18 years of age with esophageal or gastric cancer, who are living in Southern Sweden, and who are planned to undergo curative surgery treatment at Skåne University Hospital. n=100 (anticipated)
  Interventions: Other: evidence-based individualized rehabilitation
- Historical control group: The historical control group consists of patients, living in Southern Sweden, who underwent esophageal or gastric cancer surgery between 2013 - 2021 at Skåne University Hospital. n=100 (anticipated)

INTERVENTIONS:
Other: evidence-based individualized rehabilitation — The experimental group will receive structured individualized assessment based on physical, psychological or social needs and will be offered evidence-based interventions to promote rehabilitation and recovery.
  Groups: Experimental group

SUMMARY:
This study aims to develop and evaluate a model for systematic and evidence-based cancer rehabilitation for people with esophageal and gastric cancer to provide conditions for a better quality of life and fewer cancer-related symptoms.

DETAILED DESCRIPTION:
Sweden has had a National Cancer Rehabilitation Programme since 2014. This emphasises that all people with cancer have the right to individualised rehabilitation and that the contact nurse has an important role to play in identifying needs and ensuring evidence-based interventions throughout the cancer process to promote rehabilitation. The needs for optimised rehabilitation vary according to several parameters such as the person's personal circumstances and preferences, social support and type of cancer disease.

Despite this and a growing number evidence within this area cancer rehabilitation is often not integrated in clinical care. The current cancer care focuses on medical and treatment related interventions. It is a challenge for health services to find models to identify and meet the increased need for cancer rehabilitation in a systematic and structured way throughout the cancer process, based on the specific needs of each individual. This study aims to develop and evaluate a model for systematic and evidence-based cancer rehabilitation for people with esophageal and gastric cancer to provide conditions for a better quality of life and fewer cancer-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* esophageal or gastric cancer
* living in Southern Sweden (Skåne)
* are planned to undergo curative surgerytreatment at Skåne University Hospital.

Exclusion Criteria:

* unable to communicate in the Swedish language
* suffering from a cognitive impairment that poses a barrier for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: *patients over 18 years of age with esophageal or gastric cancer, who are living in Southern Sweden (Skåne), and are planned to undergo or has undergone curative surgerytreatment at Skåne University Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
General Quality of life | Instrument will be answered by the patient at baseline (at treatment decision)
  The instrument QLQ-C30 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measures quality of life. The instrument has a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit 4=very much). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items. All of the scales and single-item measures in score from 0-100. A high scale score represents a higher response level. A high score for functional scale represents a high/healthy level of functioning. A high score for global health status/QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.
General Quality of life | Instrument will be answered by the patient at approximately 1 week preoperative
  The instrument QLQ-C30 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measures quality of life. The instrument has a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit 4=very much). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items. All of the scales and single-item measures in score from 0-100. A high scale score represents a higher response level. A high score for functional scale represents a high/healthy level of functioning. A high score for global health status/QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.
General Quality of life | Instrument will be answered by the patient after surgery at 6 months postoperative
  The instrument QLQ-C30 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measures quality of life. The instrument has a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit 4=very much). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items. All of the scales and single-item measures in score from 0-100. A high scale score represents a higher response level. A high score for functional scale represents a high/healthy level of functioning. A high score for global health status/QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.
General Quality of life | Instrument will be answered by the patient after surgery at 12 months postoperative
  The instrument QLQ-C30 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measures quality of life. The instrument has a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit 4=very much). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items. All of the scales and single-item measures in score from 0-100. A high scale score represents a higher response level. A high score for functional scale represents a high/healthy level of functioning. A high score for global health status/QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.

SECONDARY OUTCOMES:
Esophageal and gastric cancer specific Quality of life | Instrument will be answered by the patient at baseline (at treatment decision)
  The instrument QLQ-OG25 is developed by the EORTC and measures diagnose specific quality of life. The instrument hast a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). The scoring approach for this instrument is identical in principle to that used for the scales/items of the EORTC-QLQ-C30.
Esophageal and gastric cancer specific Quality of life | Instrument will be answered by the patient at approximately 1 week preoperative
  The instrument QLQ-OG25 is developed by the EORTC and measures diagnose specific quality of life. The instrument hast a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). The scoring approach for this instrument is identical in principle to that used for the scales/items of the EORTC-QLQ-C30.
Esophageal and gastric cancer specific Quality of life | Instrument will be answered by the patient after surgery at 6 months postoperative
  The instrument QLQ-OG25 is developed by the EORTC and measures diagnose specific quality of life. The instrument hast a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). The scoring approach for this instrument is identical in principle to that used for the scales/items of the EORTC-QLQ-C30.
Esophageal and gastric cancer specific Quality of life | Instrument will be answered by the patient after surgery at 12 months postoperative
  The instrument QLQ-OG25 is developed by the EORTC and measures diagnose specific quality of life. The instrument hast a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). The scoring approach for this instrument is identical in principle to that used for the scales/items of the EORTC-QLQ-C30.
Information needs | Instrument will be answered by the patient at baseline (at treatment decision)
  The INFO-26 instrument is developed by the EORTC and measures the patients perception of information received. The response format is a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) in all items except four which has a two point scale (Yes/No).
Information needs | Instrument will be answered by the patient at approximately 1 week preoperative
  The INFO-26 instrument is developed by the EORTC and measures the patients perception of information received. The response format is a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) in all items except four which has a two point scale (Yes/No).
Information needs | Instrument will be answered by the patient after surgery at 6 months postoperative
  The INFO-26 instrument is developed by the EORTC and measures the patients perception of information received. The response format is a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) in all items except four which has a two point scale (Yes/No).
Information needs | Instrument will be answered by the patient after surgery at 12 months postoperative.
  The INFO-26 instrument is developed by the EORTC and measures the patients perception of information received. The response format is a four-point Likert scale (1=not at all, 2=a little, 3=quite a bit, 4=very much) in all items except four which has a two point scale (Yes/No).
International Physical Activity Questionnaire | Instrument will be answered by the patient at baseline (at treatment decision)
  The instrument IPAQ will be used to measure physical activity trough 5 questions on level of physical activity and time spent on physical activity. The IPAQ short form asks about three specific types of activities which are assessed in walking, moderate-intensity activities and vigorous-intensity activities. The instrument provides separate scores (duration and frequency) on the three types of activity.
International Physical Activity Questionnaire | Instrument will be answered by the patient at approximately 1 week preoperative
  The instrument IPAQ will be used to measure physical activity trough 5 questions on level of physical activity and time spent on physical activity. The IPAQ short form asks about three specific types of activities which are assessed in walking, moderate-intensity activities and vigorous-intensity activities. The instrument provides separate scores (duration and frequency) on the three types of activity.
International Physical Activity Questionnaire | Instrument will be answered by the patient after surgery at 6 months postoperative
  The instrument IPAQ will be used to measure physical activity trough 5 questions on level of physical activity and time spent on physical activity. The IPAQ short form asks about three specific types of activities which are assessed in walking, moderate-intensity activities and vigorous-intensity activities. The instrument provides separate scores (duration and frequency) on the three types of activity.
International Physical Activity Questionnaire | Instrument will be answered by the patient after surgery at 12 months postoperative
  The instrument IPAQ will be used to measure physical activity trough 5 questions on level of physical activity and time spent on physical activity. The IPAQ short form asks about three specific types of activities which are assessed in walking, moderate-intensity activities and vigorous-intensity activities. The instrument provides separate scores (duration and frequency) on the three types of activity.
Hospital Anxiety and Depression Scale | Instrument will be answered by the patient at baseline (at treatment decision)
  HADS will be used to measure the patients level of anxiety and depression. HADS is a 14-item scale with items for anxiety and depression subscales. Each item is rated on a 4-point Likert scale (ranging from 0=not at all, to 3=yes definitely) for a total score from 0-21 for each subscale. A higher score indicates higher levels of anxiety or depression.
Hospital Anxiety and Depression Scale | Instrument will be answered by the patient at approximately 1 week preoperative
  HADS will be used to measure the patients level of anxiety and depression. HADS is a 14-item scale with items for anxiety and depression subscales. Each item is rated on a 4-point Likert scale (ranging from 0=not at all, to 3=yes definitely) for a total score from 0-21 for each subscale. A higher score indicates higher levels of anxiety or depression.
Hospital Anxiety and Depression Scale | Instrument will be answered by the patient after surgery at 6 months postoperative
  HADS will be used to measure the patients level of anxiety and depression. HADS is a 14-item scale with items for anxiety and depression subscales. Each item is rated on a 4-point Likert scale (ranging from 0=not at all, to 3=yes definitely) for a total score from 0-21 for each subscale. A higher score indicates higher levels of anxiety or depression.
Hospital Anxiety and Depression Scale | Instrument will be answered by the patient after surgery at 12 months postoperative
  HADS will be used to measure the patients level of anxiety and depression. HADS is a 14-item scale with items for anxiety and depression subscales. Each item is rated on a 4-point Likert scale (ranging from 0=not at all, to 3=yes definitely) for a total score from 0-21 for each subscale. A higher score indicates higher levels of anxiety or depression.
Assessment of Survivorship Concerns | Instrument will be answered by the patient at baseline (at treatment decision)
  ASC will be used to measure the patients worry about cancer and worry about health trough 5 questions ranging from 1-4. Higher scores indicates greater worry.
Assessment of Survivorship Concerns | Instrument will be answered by the patient at approximately 1 week preoperative
  ASC will be used to measure the patients worry about cancer and worry about health trough 5 questions ranging from 1-4. Higher scores indicates greater worry.
Assessment of Survivorship Concerns | Instrument will be answered by the patient after surgery at 6 months postoperative
  ASC will be used to measure the patients worry about cancer and worry about health trough 5 questions ranging from 1-4. Higher scores indicates greater worry.
Assessment of Survivorship Concerns | Instrument will be answered by the patient after surgery at 12 months postoperative
  ASC will be used to measure the patients worry about cancer and worry about health trough 5 questions ranging from 1-4. Higher scores indicates greater worry.
Resilience | Instrument will be answered by the patient at baseline (at treatment decision)
  Connor-Davidsson Resilience Scale (CD-RISC) will be used to measure patients resilience trough 10 questions ranging from 0-4 Lower scores indicate more problems.
Resilience | Instrument will be answered by the patient at approximately 1 week preoperative
  Connor-Davidsson Resilience Scale (CD-RISC) will be used to measure patients resilience trough 10 questions ranging from 0-4 Lower scores indicate more problems.
Resilience | Instrument will be answered by the patientafter surgery at 6 months postoperative
  Connor-Davidsson Resilience Scale (CD-RISC) will be used to measure patients resilience trough 10 questions ranging from 0-4 Lower scores indicate more problems.
Resilience | Instrument will be answered by the patient after surgery at 12 months postoperative
  Connor-Davidsson Resilience Scale (CD-RISC) will be used to measure patients resilience trough 10 questions ranging from 0-4 Lower scores indicate more problems.
Assessment of rehabilitation needs. | Instrument will be answered by the patient at baseline (at treatment decision)
  Assessment of rehabilitation needs will be used to measure patients rehabilitation needs. A 4 point Likert scale which ranges from "no problem" to "very troublesome problem" . Higher scores indicate more problems.
Assessment of rehabilitation needs. | Instrument will be answered by the patient at approximately 1 week preoperative
  Higher scores indicate more problems.
Assessment of rehabilitation needs. | Instrument will be answered by the patient after surgery at 6 months postoperative
  Higher scores indicate more problems.
Assessment of rehabilitation needs. | Instrument will be answered by the patient after surgery at 12 months postoperative
  Higher scores indicate more problems.
Psychological Distress | Instrument will be answered by the patient at baseline (at treatment decision)
  Psychological Distress is measured by the "Distress thermometer" and will be used to measure level of distress. A scale from 0 = no distress to 10 = high distress. Higher scores indicate greater distress.
Psychological Distress | Instrument will be answered by the patient at approximately 1 week preoperative.
  Psychological Distress is measured by the "Distress thermometer" and will be used to measure level of distress. A scale from 0 = no distress to 10 = high distress. Higher scores indicate greater distress.
Psychological Distress | Instrument will be answered by the patient after surgery at 6 months postoperative.
  Psychological Distress is measured by the "Distress thermometer" and will be used to measure level of distress. A scale from 0 = no distress to 10 = high distress. Higher scores indicate greater distress.
Psychological Distress | Instrument will be answered by the patient after surgery at 12 months postoperative.
  Psychological Distress is measured by the "Distress thermometer" and will be used to measure level of distress. A scale from 0 = no distress to 10 = high distress. Higher scores indicate greater distress.
Sickness absence/work | Instrument will be answered by the patient at baseline (at treatment decision).
  Sickness abscens and to which extent the patient work will be measured by single items concerning this area.
Sickness absence/work | Instrument will be answered by the patient at approximately 1 week preoperative.
  Sickness abscens and to which extent the patient work will be measured by single items concerning this area.
Sickness absence/work | Instrument will be answered by the patient after surgery at 6 months postoperative.
  Sickness abscens and to which extent the patient work will be measured by single items concerning this area.
Sickness absence/work | Instrument will be answered by the patient after surgery at 12 months postoperative.
  Sickness abscens and to which extent the patient work will be measured by single items concerning this area.
Physical activity | Single item question will be answered by the patient at baseline (at treatment decision).
  Single item question concerning amount of hours physical activity per day.
Physical activity | Single item question will be answered by the patient at approximately 1 week preoperative.
  Single item question concerning amount of hours physical activity per day.
Physical activity | Single item question will be answered by the patient after surgery at 6 months postoperative.
  Single item question concerning amount of hours physical activity per day.
Physical activity | Single item question will be answered by the patient after surgery at 12 months postoperative.
  Single item question concerning amount of hours physical activity per day.
Alcohol use | Single item questions will be answered by the patient at baseline (at treatment decision).
  Single item questions concerning alcohol use.
Alcohol use | Single item questions will be answered by the patient at approximately 1 week preoperative.
  Single item questions concerning alcohol use.
Alcohol use | Single item questions will be answered by the patient after surgery at 6 months postoperative.
  Single item questions concerning alcohol use.
Alcohol use | Single item questions will be answered by the patient after surgery at 12 months postoperative.
  Single item questions concerning alcohol use.
Tobacco use | Single item questions will be answered by the patient at baseline (at treatment decision).
  Single item questions concerning tobacco use.
Tobacco use | Single item questions will be answered by the patient at approximately 1 week preoperative.
  Single item questions concerning tobacco use.
Tobacco use | Single item questions will be answered by the patient after surgery at 6 months postoperative.
  Single item questions concerning tobacco use.
Tobacco use | Single item questions will be answered by the patient after surgery at 12 months postoperative.
  Single item questions concerning tobacco use.
Height | Single item question will be answered by the patient at baseline (at treatment decision).
  Single item question concerning height in meters.
Weight | Single item question will be answered by the patient at baseline (at treatment decision).
  Single item question concerning weight in kilograms.
Weight | Single item question will be answered by the patient at approximately 1 week preoperative.
  Single item question concerning weight in kilograms.
Weight | Single item question will be answered by the patient after surgery at 6 months postoperative.
  Single item question concerning weight in kilograms.
Weight | Single item question will be answered by the patient after surgery at 12 months postoperative.
  Single item question concerning weight in kilograms.
Body Mass Index (BMI) | Instrument will be answered by the patient after surgery at baseline (at treatment decision).
  Weight and height will be combined to report BMI in kg/m^2.
Body Mass Index (BMI) | Instrument will be answered by the patient at approximately 1 week preoperative.
  Weight and height will be combined to report BMI in kg/m^2.
Body Mass Index (BMI) | Instrument will be answered by the patient after surgery at 6 months postoperative.
  Weight and height will be combined to report BMI in kg/m^2.
Body Mass Index (BMI) | Instrument will be answered by the patient after surgery at 12 months postoperative.
  Weight and height will be combined to report BMI in kg/m^2.
Dysphagia | Instrument will be answered by the patient at baseline (at treatment decision).
  Dysphagia will be measured by a single item concerning how it works to swallow for the patient and it ranges from 0-4 (0=no dysphagia to 4=total dysphagia) Higher scores indicate more difficulties swallowing.
Dysphagia | Instrument will be answered by the patient at approximately 1 week preoperative.
  Dysphagia will be measured by a single item concerning how it works to swallow for the patient and it ranges from 0-4 (0=no dysphagia to 4=total dysphagia) Higher scores indicate more difficulties swallowing.
Dysphagia | Instrument will be answered by the patient after surgery at 6 months postoperative.
  Dysphagia will be measured by a single item concerning how it works to swallow for the patient and it ranges from 0-4 (0=no dysphagia to 4=total dysphagia) Higher scores indicate more difficulties swallowing.
Dysphagia | Instrument will be answered by the patient after surgery at 12 months postoperative.
  Dysphagia will be measured by a single item concerning how it works to swallow for the patient and it ranges from 0-4 (0=no dysphagia to 4=total dysphagia) Higher scores indicate more difficulties swallowing.
Rehabilitation process | Instrument will be answered by the patient at baseline (at treatment decision).
  Questions about the rehabilitation process will be measured by single items concerning this area.
Rehabilitation process | Instrument will be answered by the patient at approximately 1 week preoperative.
  Questions about the rehabilitation process will be measured by single items concerning this area.
Rehabilitation process | Instrument will be answered by the patient after surgery at 6 months postoperative.
  Questions about the rehabilitation process will be measured by single items concerning this area.
Rehabilitation process | Instrument will be answered by the patient after surgery at 12 months postoperative.
  Questions about the rehabilitation process will be measured by single items concerning this area.

OTHER OUTCOMES:
Demographics | The data will be collected 12 months after surgery.
  Demographic details will be collected from participants via NREV (Swedish national quality registry for esophageal and gastric cancer). There are no scales, only quality registry data.This data includes gender,cancerdiagnosis, tumourstage, comorbidity according to ASA, surgerydate, postoperative tumourstage.
Overall survival | Up to 1 year after surgery
  Overall survival will be collected from participants via NREV (Swedish national quality registry for esophageal and gastric cancer). There are no scales, only quality registry data.
Incidence and severity of general complications | Up to 30 days postoperative
  Incidence rate and severity of general complication according to Clavien-Dindo classification. Genereal complications will be collected from participants via NREV (Swedish national quality registry for esophageal and gastric cancer).
Change of level of care | Up to 30 days postoperative
  Incidence rate of change of level of care in the context of postoperative care will be collected from participants via NREV (Swedish national quality registry for esophageal and gastric cancer).
Length of stay | from the day before surgery to discharge from the hospital
  Length of stay at the hospital will be collected from participants via NREV (Swedish national quality registry for esophageal and gastric cancer). Will be measured in number of days.
Rate of re-admission | Up to 30 days postoperative
  The rate of re-admission up to 30 days postoperative will be collected via NREV (Swedish national quality registry for esophageal and gastric cancer).
Discharge destination | The data will be collected 12 months postoperative
  Postoperative discharge destination (i.e if the patients goes home or to another care unit after discharge) will be collected via NREV (Swedish national quality registry for esophageal and gastric cancer)

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No